CLINICAL TRIAL: NCT01214876
Title: Correlating Protection Against Malaria With Serum Profiles Against Plasmodium Falciparum Antigen Repertoires
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other); Medical Biotech Laboratories (Unknown); University Of Perugia (Other); Imperial College London (Other); Microtest Matrices Ltd (Unknown)
Responsible Party: Teun Bousema, London School of Hygiene & Tropical Medicine
Other Study IDs: FIGHTMAL
Record Dates: First submitted 2010-10-04; First posted 2010-10-05 (Estimated); Last update posted 2011-03-04 (Estimated); Status verified 2010-08

CONDITIONS: Malaria; Schistosomiasis; Hiv Infection
MeSH Terms: conditions — Malaria; Schistosomiasis; HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma samples Human DNA samples Parasite DNA samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Children 1-5 years old
- Children 6-10 years old
- Adults 25 years and above

SUMMARY:
A longitudinal study on immune responses in relation to protection against clinical malaria episodes will be conducted in Apac District, Uganda. Three cohorts will be recruited: children 1 to 5 years of age (n=250), children 6 to 10 years of age (n=125) and adults 25 and above (n=125). After finger prick sampling (~300µL) and examination at enrolment, participants will be followed up for one year. Follow-up will include fortnightly active case detection and three-monthly cross-sectional surveys. Clinical malaria attacks and the associated clinical and parasitological parameters will be related to immunological profiles determined utilizing a protein microarray as a capture substratum to profile the humoral immune response against a vast number of parasite antigens.

For individuals who experience a clinical malaria attack or who are diagnosed with high density parasitaemia (≥15,000 parasites/µL) during cross-sectional surveys, a 5mL blood sample is obtained to determine the diversity of parasite antigens in the population in relation to antigen recognition in the cohort.

ELIGIBILITY:
Inclusion Criteria:

* age 1-5 years, 6-10 years or 25 yearsand above
* written informed consent must be given
* the individual must have been resident of the area since birth or for a minimum period of two years
* the individual must be willing to submit required information and to participate in repeated sampling (total blood volume ~2.5 mL over a period of 12 months)
* Absence of danger signs (as defined by WHO) or clinical features of AIDS. An HIV-test will be offered to all participants at enrolment and completion of the study.

Exclusion Criteria:

* unwillingness to sign consent form
* unwillingness to reside in the study area during the follow-up period

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Randomly selected individuals living in Abedi, Apac District, Uganda.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2010-08; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Immune correlates of protection against clinical malaria episodes with plasmodium falciparum
  IMMUNE RESPONSES: protein array.
  CLINICAL MALARIA EPISODES: (reported) fever with i) P. falciparum parasites; ii) ... at a density >=5,000 parasites/ul; iii) ... at a density >=10,000 parasites/ul IMMUNOLOGICALLY PROTECTED INDIVIDUALS: parasitaemic during follow-up without reporting to the health facility with indicators of a clinical malaria episode

SECONDARY OUTCOMES:
Geographical patterns in malaria morbidity
  Households are geo-located by GPS and hotspots of malaria transmission will be determined and related to serological profiles.
Asymptomatic parasite carriage and immune responses in different age-groups exposed to intense malaria transmission
  ASYMPTOMATIC PARASITE CARRIAGE will be confirmed by microscopy and PCR.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Biotech Laboratories, Kampala, Uganda